CLINICAL TRIAL: NCT07078110
Title: Comparative Evaluation of Clinical Performance of Bulk-Fill Composites With Incrementally Layered Conventional Composites: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Clinical Performance of Bulk-Fill Composites With Incrementally Layered Conventional Composites
Acronym: ILCVSBFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Dental College (Other)
Responsible Party: Principal Investigator, Maliha Hameed, Assistant Professor Paedodontics, Fatima Jinnah Dental College
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FEB-2017-OPR02
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Sensitivity; Anatomic Form of the Restoration; Colour Match of the Restoration; Marginal Discolouration; Marginal Adaptation; Secondary Caries; Retention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Control Group:
  Group I (Incremental Technique):
  Applied in 2 mm incremental layers, light-cured for 40 seconds per increment Material: Filtek Z250 (3M ESPE, USA)
  Interventions: Procedure: Material: Filtek Z250 (3M ESPE, USA)
- Experimental group (Active Comparator): Group II (Bulk-Fill Technique):
  Applied in a single increment (up to 4 mm) and light-cured for 40 seconds. Material: Filtek Bulk-Fill Restorative (FBF), 3M ESPE, USA
  Interventions: Procedure: Material: Filtek Bulk-Fill Restorative (FBF), 3M ESPE, USA

INTERVENTIONS:
Procedure: Material: Filtek Z250 (3M ESPE, USA) — Group I (Incremental Technique):
  Material: Filtek Z250 (3M ESPE, USA) Applied in 2 mm incremental layers, light-cured for 40 seconds per increment.
  Arms: Control Group
Procedure: Material: Filtek Bulk-Fill Restorative (FBF), 3M ESPE, USA — Group II (Bulk-Fill Technique):
  Material: Filtek Bulk-Fill Restorative (FBF), 3M ESPE, USA Applied in a single increment (up to 4 mm) and light-cured for 40 seconds.
  Arms: Experimental group

SUMMARY:
This study aimed to compare the clinical effectiveness of bulk-fill composites with conventionally layered incremental composites in Class I cavities using modified USPHS criteria. Fifty patients were selected based on sample size calculations. Each patient received two restorations, one from each group. Group I received incremental layering composite restorations, while Group II received bulk-fill composite restorations. Group I restorations were placed on the right side, and Group II restorations were placed on the left side. A single trained operator placed all restorations. After one year, the restorations were evaluated using modified USPHS criteria. Periapical radiographs were taken, and postoperative sensitivity was assessed using cold testing (ethyl chloride spray), with pain responses recorded using the Visual Analogue Scale.

DETAILED DESCRIPTION:
This study aimed to compare the clinical effectiveness of bulk-fill composites with conventionally layered incremental composites in Class I cavities using modified USPHS criteria. Patients aged 15 to 50 years of either gender visiting Fatima Jinnah Dental College and Hospital OPD who fulfilled the inclusion criteria (vital first and second molar teeth with Class I cavities having a depth of 3-4mm) were recruited in the study from July 2021 to January 2023. Fifty patients were selected based on sample size calculations. Each patient received two restorations, one from each group. Group I received incremental layering composite restorations, while Group II received bulk-fill composite restorations. Group I restorations were placed on the right side, and Group II restorations were placed on the left side. A single trained operator placed all restorations. After one year, the restorations were evaluated using modified USPHS criteria. Periapical radiographs were taken, and postoperative sensitivity was assessed using cold testing (ethyl chloride spray), with pain responses recorded using the Visual Analogue Scale.

Eligibility Criteria:

Inclusion Criteria:

Patients aged 15 to 50 years, of either gender. Visiting Fatima Jinnah Dental College and Hospital OPD. Vital first and second molar teeth with Class I cavities, 3-4 mm in depth.

Exclusion Criteria:

Patients with xerostomia or bruxism (assessed via medical history). Teeth with irreversible pulpitis or necrotic pulps. Previously restored or periodontally compromised teeth.

Confounding Variables:

Confounding factors like xerostomia and bruxism were excluded. Factors like smoking and soft drink consumption were considered during analysis.

Preoperative Assessment Electric pulp tester was used to evaluate tooth vitality. Adjacent tissues were clinically examined. Baseline data included age, sex, tooth treated, and caries depth.

Operative Procedure Local anesthesia was administered using 2% lidocaine (1.8 ml cartridge). Rubber dam isolation was employed for moisture control. Cavity preparation was done using a straight fissure bur in a high-speed handpiece.

Carious dentin was removed using a spoon excavator or slow-speed tungsten carbide bur.

Etching followed by application of 3M Singlebond Universal adhesive for 35 seconds, gently air-dried, then light-cured for 20 seconds.

Restoration Groups

Each participant received two restorations-one from each group-to allow for intra-individual comparison:

Group I (Incremental Technique):

Material: Filtek Z250 (3M ESPE, USA) Applied in 2 mm incremental layers, light-cured for 40 seconds per increment.

Group II (Bulk-Fill Technique):

Material: Filtek Bulk-Fill Restorative (FBF), 3M ESPE, USA Applied in a single increment (up to 4 mm) and light-cured for 40 seconds.

Group I restorations were placed on the right side, and Group II on the left side. All restorations were placed by a single trained operator over 6 months. The participants were blinded to the type of restoration used.

Follow-Up and Evaluation Restorations were evaluated 1 year post-placement by a principal investigator under a dental operating light using flat-surfaced mouth mirrors and dental explorers.

Evaluation followed modified USPHS criteria, assessing:

Anatomic form Color match Marginal discoloration Marginal adaptation Secondary caries Retention

STATISTICAL ANALYSIS:

Descriptive statistics and post-stratification Chi-square tests were performed.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Patients aged 15 to 50 years, of either gender. Visiting Fatima Jinnah Dental College and Hospital OPD. Vital first and second molar teeth with Class I cavities, 3-4 mm in depth.

Exclusion Criteria:

Patients with xerostomia or bruxism (assessed via medical history). Teeth with irreversible pulpitis or necrotic pulps. Previously restored or periodontally compromised teeth.

Confounding Variables:

Confounding factors like xerostomia and bruxism were excluded. Factors like smoking and soft drink consumption were considered during analysis.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Postoperative senstivity | One year
  Postoperative sensitivity was assessed using ethyl chloride spray and scored using the Visual Analogue Scale (VAS):
  0 = No pain 1-3 cm = Mild pain 4-6 cm = Moderate pain 7-10 cm = Severe pain

SECONDARY OUTCOMES:
Anatomic form | One year
  Assesses the restoration's shape and how well it conforms to the natural contours of the tooth.
  Alfa: Continuous Bravo: Slight discontinuity, clinically acceptable Charlie: Discontinuous, failure
Colour match | One year
  Evaluates how well the restoration blends with the surrounding natural tooth color.
  Alfa: Matches tooth Bravo: Acceptable mismatch Charlie: Unacceptable mismatch
Marginal discolouration | One year
  Examines the presence of any dark lines or discoloration along the margins of the restoration.
  Alfa: No discoloration Bravo: Discoloration without Charlie: Discoloration with penetration in pulpal direction
Marginal Adaptation | One year
  Evaluates the fit of the restoration at the margins, looking for any gaps or discrepancies.
  Alfa: Closely adapted, no visible crevice Bravo: Visible crevice, explorer will penetrate Charlie: Crevice in which dentin is exposed
Secondary caries | One year
  Examines the presence of new decay around the restoration, indicating potential failure.
  Alfa: No caries present Charlie: Caries present
Retention | One year
  Assesses whether the restoration remains firmly in place and hasn't fractured or dislodged.
  Alfa: No loss of restorative material Charlie: Any loss of restorative material

CONTACTS AND LOCATIONS:
Overall Officials: Dr Maliha Naveed Assistant Professor, Principal Investigator — Bahria University Medical & Dental College
Locations (1):
- Fatima Jinnah Dental College, Hospital Karachi Pakistan, Karachi, Pakistan

REFERENCES:
- [Derived] Naveed M, Ahmed MA, Syed AUY, Saqib M, Ali M, Jouhar R, Faheemuddin M, Umer MF. Comparative evaluation of clinical performance of bulk-fill composites with incrementally layered conventional composites. BMC Oral Health. 2025 Dec 5;26(1):55. doi: 10.1186/s12903-025-07453-6. PMID 41345621